CLINICAL TRIAL: NCT02503332
Title: A Phase II, Multicenter, Randomized, Single-Masked, Sham-Controlled Study of Safety, Tolerability and Evidence of Activity of Intravitreal APL-2 Therapy in Patients With Geographic Atrophy (GA)
Brief Title: Study of Pegcetacoplan (APL-2) Therapy in Patients With Geographic Atrophy
Acronym: FILLY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: POT-CP121614
Record Dates: First submitted 2015-07-14; First posted 2015-07-20 (Estimated); Results first posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy | interventions — pegcetacoplan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pegcetacoplan 15 mg/100 µL Monthly for 12 months (Experimental): A single dose of 15 mg pegcetacoplan/100 µL will be administered via intravitreal injection in this study. Subjects will receive an injection every month for 12 consecutive months.
  Interventions: Drug: Pegcetacoplan
- Pegcetacoplan 15 mg/100 µL EOM for 12 months (Experimental): A single dose of 15 mg pegcetacoplan/100 µL will be administered via intravitreal injection in this study. Subjects will receive an injection every other month (EOM) for 12 consecutive months.
  Interventions: Drug: Pegcetacoplan
- Sham Monthly for 12 months (Sham Comparator): Subjects will receive a Sham procedure every month for 12 consecutive months.
  Interventions: Other: Sham Procedure
- Sham EOM for 12 months (Sham Comparator): Subjects will receive a Sham procedure every other month (EOM) for 12 consecutive months.
  Interventions: Other: Sham Procedure

INTERVENTIONS:
Drug: Pegcetacoplan
  Other Names: APL-2
  Arms: Pegcetacoplan 15 mg/100 µL EOM for 12 months; Pegcetacoplan 15 mg/100 µL Monthly for 12 months
Other: Sham Procedure
  Arms: Sham EOM for 12 months; Sham Monthly for 12 months

SUMMARY:
The primary objectives of the study are to assess the safety, tolerability and evidence of activity of multiple intravitreal (IVT) injections of pegcetacoplan in subjects with Geographic Atrophy associated with Age-Related Macular Degeneration (AMD).

DETAILED DESCRIPTION:
This is a Phase II, prospective, multicenter, randomized, single-masked, sham-controlled study to assess the safety, tolerability and evidence of activity of multiple IVT injections of pegcetacoplan in subjects with GA secondary to Age-Related Macular Degeneration.

The study will randomize approximately 240 subjects to obtain at least 200 evaluable subjects across 40 multinational sites.

Subjects will be randomized in a 2:2:1:1 manner to receive pegcetacoplan Monthly (AM), pegcetacoplan Every-Other-Month (AEOM), Sham injection Monthly (SM) or Sham injection Every-Other-Month (SEOM), respectively.

All subjects will return to the clinical site on Day 7 to assess acute safety after the first injection. After that, subjects in the monthly groups will return to the clinical site for additional pegcetacoplan (or Sham) injections and study procedures every month until Month 12. Subjects in the Every-Other-Month groups will return to the clinical site for additional pegcetacoplan (or Sham) injections and study procedures every two months until Month 12. All subjects will return for follow-up visits on Months 15 and 18 (3 and 6 months after last injection, respectively).

ELIGIBILITY:
Inclusion Criteria: Unless specified otherwise, ocular specific inclusion criteria apply to the study eye only.

1. Male or Female.
2. Age greater than or equal to 50 years.
3. BCVA of 20/320 (Snellen equivalent) or better using ETDRS charts.
4. Diagnosis of GA of the macula secondary to age-related macular degeneration, confirmed within 14 days prior to randomization by the central reading center (CRC) using Fundus Autofluorescence (FAF) images, as well as the following criteria:

   1. Total GA area must be ≥ 2.5 and ≤ 17.5 mm2 (1 and 7 disk areas [DA] respectively), determined by screening images of FAF.
   2. If GA is multifocal, at least one focal lesion must be ≥ 1.25 mm2 (0.5 DA).
   3. GA can be completely visualized on the macula centered image.
   4. GA must be able to be photographed in its entirety.
   5. GA must be able to be measured separately from any areas of peripapillary atrophy as assessed by the CRC.
   6. Presence of any pattern of hyperautofluorescence in the junctional zone of GA. Absence of hyperautoflouorescence (i.e. pattern = none) is exclusionary. See Holz et al. 2007.1
5. Female subjects must be:

   1. Women of non-child-bearing potential (WONCBP), or
   2. Women of child-bearing potential (WOCBP) with a negative pregnancy test at screening and must agree to use protocol defined methods of contraception for the duration of the study.
6. Males with female partners of child-bearing potential must agree to use protocol defined methods of contraception and agree to refrain from donating sperm for the duration of the study.
7. Willing and able to give informed consent.

Exclusion Criteria: Unless specified otherwise, ocular specific inclusion criteria apply to the study eye only.

1. GA due to causes other than AMD such as Stargardt disease, cone rod dystrophy or toxic maculopathies like plaquenil maculopathy.
2. Spherical equivalent of the refractive error demonstrating > 6 diopters of myopia or an axial length >26 mm.
3. Any history or current evidence of exudative ("wet") AMD including any evidence of retinal pigment epithelium rips or evidence of neovascularization anywhere in the retina based on fluorescein angiogram as assessed by the CRC.
4. Retinal disease other than AMD; however, benign conditions of the vitreous or peripheral retina are not exclusionary (i.e. pavingstone degeneration).
5. Any ophthalmologic condition that reduces the clarity of the media and that, in the opinion of the Investigator interferes with ophthalmologic examination (e.g. advanced cataract or corneal abnormalities).
6. Any ophthalmologic condition that prevents adequate imaging of the retina judged by the site or CRC.
7. Intraocular surgery (including lens replacement surgery) within 3 months prior to randomization.
8. Aphakia or absence of the posterior capsule. Previous violation of the posterior capsule is also excluded unless it occurred as a result of yttrium aluminum garnet (YAG) laser posterior capsulotomy in association with prior posterior chamber intraocular lens implantation and at least 60 days prior to Day 0.
9. Any ophthalmic condition that may require surgery during the study period.
10. Any contraindication to IVT injection including current ocular or periocular infection.
11. History of uveitis or endophthalmitis.
12. History of IVT injection at any time.
13. Participation in another interventional clinical study, or use of any experimental treatment for AMD or any other investigational new drug within 6 weeks or 5 half-lives of the active (whichever is longer) prior to the start of study treatment. Note: clinical trials solely involving observation, over-the-counter vitamins, supplements, or diets are not exclusionary.
14. Medical or psychiatric conditions that, in the opinion of the investigator, make consistent follow-up over the treatment period unlikely, or in general a poor medical risk because of other systemic diseases or active uncontrolled infections.
15. Any screening laboratory value (hematology, serum chemistry or urinalysis) that in the opinion of the Investigator is clinically significant and not suitable for study participation.
16. Hypersensitivity to fluorescein.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2018-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Grossi, MD PhD, Study Director — Apellis Pharmaceuticals, Inc.
Locations (46):
- United States (35):
  - Retina Speciality Institute, Mobile, Alabama
  - Retinal Research Institute, Phoenix, Arizona
  - Retina Vitreous Asociates Mdical Goup, Beverly Hills, California
  - The Gavin Herbert Eye Institute/UC Irvine, Irvine, California
  - University of Southern California - USC Eye Institute, Los Angeles, California
  - Byers Eye Institute at Stanford, Stanford School of Medicine, Palo Alto, California
  - New England Retina Associates, New London, Connecticut
  - Florida Eye Microsurgical Institute, Inc., Boynton Beach, Florida
  - Retina Health Center, Fort Myers, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - South East Retina, Augusta, Georgia
  - Illinois Retina Associates, Harvey, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Elman Research, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Associated Retinal Consultants PC, Grand Rapids, Michigan
  - Associated Retinal Consultants, PC, Traverse City, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Eyesight Opthalmic Services PA, Portsmouth, New Hampshire
  - Vitreous Retina Macula Consultants of New York, New York, New York
  - Charlotte Eye Ear Nose and Throat Associates, Charlotte, North Carolina
  - Duke University, Duke Eye Center, Durham, North Carolina
  - Charlotte Eye Ear Nose and Throat Associates, Statesville, North Carolina
  - Cleveland Clinic Foundation/ Cole Eye Institute, Cleveland, Ohio
  - Retina Associates of Cleveland, Cleveland, Ohio
  - Mid Atlantic, Philadelphia, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Tennessee Retina, PC, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Retina Research Center, Austin, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - Retina Specialists, Plano, Texas
  - Retina Consultants of Houston (The Woodlands), The Woodlands, Texas
  - University of Utah, Salt Lake City, Utah
- Australia (9):
  - Marsden Eye Specialists, Paramatta, New South Wales
  - Save Sight Institute, Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
  - Sydney West Retina, Westmead, New South Wales
  - Hobart eye Surgeons, Hobart, Tasmania
  - Tasmanian Eye Institute, South Launceston, Tasmania
  - Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria
  - Center for Eye Research Australia, Melbourne, Victoria
  - Lions Eye Institute, Nedlands, Western Australia
- New Zealand (2):
  - Auckland Eye, Remuera, Auckland
  - Southern Eye Specialists, Merivale, Christchurch

REFERENCES:
- [Derived] Reiter GS, Lachinov D, Buhl W, Weigert G, Grechenig C, Mai J, Bogunovic H, Schmidt-Erfurth U. A Novel Management Challenge in Age-Related Macular Degeneration: Artificial Intelligence and Expert Prediction of Geographic Atrophy. Ophthalmol Retina. 2025 May;9(5):421-430. doi: 10.1016/j.oret.2024.10.029. Epub 2024 Nov 9. PMID 39522752
- [Derived] Fu DJ, Lipkova V, Liefers B, Glinton S, Faes L, McKeown A, Scheibler L, Pontikos N, Patel PJ, Zhang G, Keane PA, Balaskas K. Evaluating the Effects of C3 Inhibition on Geographic Atrophy Progression from Deep-Learning OCT Quantification: A Split-Person Study. Ophthalmol Ther. 2023 Dec;12(6):3143-3158. doi: 10.1007/s40123-023-00798-7. Epub 2023 Sep 16. PMID 37715860
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061
- [Derived] Pfau M, Schmitz-Valckenberg S, Ribeiro R, Safaei R, McKeown A, Fleckenstein M, Holz FG. Association of complement C3 inhibitor pegcetacoplan with reduced photoreceptor degeneration beyond areas of geographic atrophy. Sci Rep. 2022 Oct 25;12(1):17870. doi: 10.1038/s41598-022-22404-9. PMID 36284220
- [Derived] Vogl WD, Riedl S, Mai J, Reiter GS, Lachinov D, Bogunovic H, Schmidt-Erfurth U. Predicting Topographic Disease Progression and Treatment Response of Pegcetacoplan in Geographic Atrophy Quantified by Deep Learning. Ophthalmol Retina. 2023 Jan;7(1):4-13. doi: 10.1016/j.oret.2022.08.003. Epub 2022 Aug 7. PMID 35948209
- [Derived] Liao DS, Metlapally R, Joshi P. Pegcetacoplan treatment for geographic atrophy due to age-related macular degeneration: a plain language summary of the FILLY study. Immunotherapy. 2022 Sep;14(13):995-1006. doi: 10.2217/imt-2022-0078. Epub 2022 Jul 21. PMID 35860926
- [Derived] Nittala MG, Metlapally R, Ip M, Chakravarthy U, Holz FG, Staurenghi G, Waheed N, Velaga SB, Lindenberg S, Karamat A, Koester J, Ribeiro R, Sadda S. Association of Pegcetacoplan With Progression of Incomplete Retinal Pigment Epithelium and Outer Retinal Atrophy in Age-Related Macular Degeneration: A Post Hoc Analysis of the FILLY Randomized Clinical Trial. JAMA Ophthalmol. 2022 Mar 1;140(3):243-249. doi: 10.1001/jamaophthalmol.2021.6067. PMID 35113137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase II, randomized, single-masked, sham injection-controlled study in subjects with geographic atrophy (GA) secondary to age-related macular degeneration (AMD) was conducted at 47 sites (46 active) in 3 countries between 24 September 2015 and 14 July 2017 (Data cut-off date, Month 12).
Pre-assignment Details: Subjects were randomized in a 2:2:1:1 manner to receive treatment with pegcetacoplan monthly, pegcetacoplan every-other-month (EOM), sham monthly or sham EOM, respectively. A total of 246 subjects were randomized in the study.
Groups:
- Pegcetacoplan Monthly: Subjects received intravitreal (IVT) injections of pegcetacoplan 15 milligrams (mg)/100 microliters (μL) once monthly for 12 months.
- Pegcetacoplan EOM: Subjects received IVT injections of pegcetacoplan 15 mg/100 μL EOM for 12 months.
- Sham Monthly: Subjects received sham injections once monthly for 12 months. The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
- Sham EOM: Subjects received sham injections EOM for 12 months. The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
Period: Overall Study
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Monthly | Sham EOM
Started | 86 | 79 | 41 | 40
Completed (Completed treatment.) | 52 | 60 | 33 | 36
Not Completed | 34 | 19 | 8 | 4
Not completed — Adverse Event | 17 | 5 | 3 | 1
Not completed — Investigator's Decision | 5 | 1 | 0 | 0
Not completed — Sponsor's Decision | 1 | 0 | 0 | 1
Not completed — Subject Request | 6 | 5 | 2 | 1
Not completed — Death | 0 | 2 | 2 | 0
Not completed — Other | 5 | 6 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) population included all randomized subjects who received at least one injection of study drug.
Groups:
- Pegcetacoplan Monthly: Subjects received IVT injections of pegcetacoplan 15 mg/100 μL once monthly for 12 months.
- Sham Pooled: Sham Monthly: Subjects received sham injections once monthly for 12 months.
  Sham EOM: Subjects received sham injections EOM for 12 months. The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
- Total: Total of all reporting groups
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled | Total
Number analyzed (Participants) | 86 | 79 | 81 | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.6 (7.51) | 81.0 (7.55) | 78.4 (7.43) | 79.7 (7.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 50 | 49 | 154
  Male | 31 | 29 | 32 | 92
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Black or African American | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 84 | 76 | 81 | 241
  Other | 0 | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 5
  Not Hispanic or Latino | 81 | 76 | 77 | 234
  Not Reported | 2 | 0 | 0 | 2
  Unknown | 1 | 2 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 12 | 11 | 12 | 35
  New Zealand | 3 | 3 | 4 | 10
  United States | 71 | 65 | 65 | 201
GA Lesion Size (fundus autofluorescence [FAF]) in the Study Eye [Mean (Standard Deviation); unit: millimeter square (mm^2)] | 8.0 (3.84) | 8.9 (4.47) | 8.2 (4.05) | 8.4 (4.12)

OUTCOME MEASURES:

1. Primary Outcome: Least Square (LS) Mean Change From Baseline in Square Root GA Lesion Size in the Study Eye at Month 12
Description: The square root GA lesion size (i.e. transformed area of GA) was measured by FAF photographs. Baseline was defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: Baseline (screening) and Month 12.
Population: The modified ITT (mITT) population included all randomized subjects who received at least one injection of study drug and had at least one visit at or after Month 2 where primary efficacy data was collected. Subjects were included in their randomized treatment group even if they received the wrong study drug.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 84 | 78 | 80
mm | 0.26 (0.025) | 0.28 (0.026) | 0.35 (0.025)

2. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs) in the Study Eye, Including by Severity
Description: A TEAE was defined as any adverse event (AE) that commenced or worsened on or after time of first study drug administration up to 60 days beyond last dose of study drug. A treatment-related TEAE was defined as a TEAE with a relationship to study drug of possibly related or probably related or not reported. Severity of TEAEs were categorized as mild; moderate; severe; life-threatening or death related to TEAE, according to Common Terminology Criteria for AEs v4.03. A TEAE of special interest (TEAESI) was defined as a TEAE of scientific and medical concern specific to pegcetacoplan, whether serious or non-serious.
Time Frame: From the time of first study drug administration (Day 1) up to Month 12 (Data cut-off date).
Population: The safety population included all randomized subjects who received at least one injection of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 86 | 79 | 81
Participants
  TEAEs | 65 | 47 | 42
  Treatment-related TEAEs | 21 | 11 | 0
  Serious TEAEs | 4 | 2 | 1
  TEAEs with mild intensity | 36 | 30 | 28
  TEAEs with moderate intensity | 23 | 14 | 11
  TEAEs with severe intensity | 6 | 3 | 3
  TEAEs with life-threatening intensity | 0 | 0 | 0
  Death related to TEAEs | 0 | 0 | 0
  TEAESIs | 5 | 4 | 0
  TEAEs leading to study/treatment discontinuation | 19 | 5 | 3

3. Secondary Outcome: LS Mean Change From Baseline in Untransformed GA Lesion Size in the Study Eye at Month 12
Description: The untransformed area of GA was measured by FAF. Baseline is defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: Baseline (Day 1) and Month 12.
Population: The mITT population included all randomized subjects who received at least one injection of study drug and had at least one visit at or after Month 2 where primary efficacy data was collected. Subjects were included in their randomized treatment group even if they received the wrong study drug.
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 84 | 78 | 80
mm^2 | 1.49 (0.161) | 1.69 (0.168) | 2.12 (0.161)

4. Secondary Outcome: LS Mean Change From Baseline in Best-Corrected Visual Acuity (BCVA) Score of the Study Eye at Month 12
Description: The BCVA letter score was determined using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. The score ranges from 0 to 100 letters, lower number indicating reduced visual acuity; a positive value of change from baseline indicates visual acuity gain and a negative value indicates visual acuity loss.
Time Frame: Baseline (Day 1) and Month 12.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ETDRS letter score
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 84 | 78 | 80
ETDRS letter score | -3.31 (1.352) | -5.78 (1.398) | -4.36 (1.364)

5. Secondary Outcome: LS Mean Change From Baseline in Low Luminance BCVA (LL-BCVA) Score in the Study Eye at Month 12
Description: The LL-BCVA was measured by placing a 2.0-log-unit neutral density filter over the best correction and having the participant read the normally illuminated ETDRS chart. The score ranges from 0 to 100 letters, lower number indicating worse vision; a positive value of change from baseline indicates visual acuity gain and a negative value indicates visual acuity loss.
Time Frame: Baseline (Day 1) and Month 12.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ETDRS letter score
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 84 | 78 | 80
ETDRS letter score | -2.73 (1.145) | -3.21 (1.184) | -0.55 (1.150)

6. Secondary Outcome: LS Mean Change From Baseline in Low Luminance VA (LL-VA) Deficit Score in the Study Eye at Month 12
Description: The LL-VA deficit score is calculated as BCVA score minus LL-BCVA score. The LL-VA deficit score ranges from 0 to 100 letters, lower number indicating worse deficit.
Time Frame: Baseline (Day 1) and Month 12.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ETDRS letter score
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 84 | 78 | 80
ETDRS letter score | -0.76 (1.382) | -2.40 (1.424) | -3.72 (1.385)

7. Secondary Outcome: LS Mean Change From Baseline in Distance of GA Lesion From the Fovea (Foveal Encroachment) in the Study Eye at Month 12
Description: The foveal encroachment in the study eye was measured by FAF. Baseline is defined as the last available, non-missing observation prior to first study drug administration.
Time Frame: Baseline (Day 1) and Month 12.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 84 | 78 | 80
mm | -0.04 (0.011) | -0.04 (0.012) | -0.06 (0.011)

8. Secondary Outcome: Number of Subjects With Any Macular Neovascularization (MNV) TEAEs in the Study Eye
Description: The number of subjects with any MNV TEAEs in the study eye was identified via clinical review of all ocular TEAEs.
Time Frame: From the time of first study drug administration (Day 1) up to Month 12 (Data cut-off date).
Population: The safety population included all randomized subjects who received at least one injection of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan Monthly | Pegcetacoplan EOM | Sham Pooled
Number analyzed (Participants) | 86 | 79 | 81
Participants | 14 | 5 | 1

ADVERSE EVENTS:
Time Frame: TEAE data is reported from the time of first study drug administration (Day 1) up to Month 12 (Data cut-off date).
Description: The safety population included all randomized subjects who received at least one injection of study drug.
  Ocular TEAEs are presented separately for the study and fellow eyes, and non-ocular (systemic) TEAEs are also presented.
Groups:
- Pegcetacoplan Monthly: Ocular Study Eye: Ocular TEAEs are summarized for the study eye for all subjects who received IVT injections of pegcetacoplan 15 mg/100 μL once monthly for 12 months.
- Pegcetacoplan EOM: Ocular Study Eye: Ocular TEAEs are summarized for the study eye for all subjects who received IVT injections of pegcetacoplan 15 mg/100 μL EOM for 12 months.
- Sham Pooled: Ocular Study Eye: Ocular TEAEs are summarized for the study eye for all subjects who randomized to sham monthly and sham EOM treatment groups.
  Sham Monthly: Subjects received sham injections once monthly for 12 months.
  Sham EOM: Subjects received sham injections EOM for 12 months. The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
- Pegcetacoplan Monthly: Ocular Fellow Eye: Ocular TEAEs are summarized for the fellow eye for all subjects who received IVT injections of pegcetacoplan 15 mg/100 μL once monthly for 12 months.
- Pegcetacoplan EOM: Ocular Fellow Eye: Ocular TEAEs are summarized for the fellow eye for all subjects who received IVT injections of pegcetacoplan 15 mg/100 μL EOM for 12 months.
- Sham Pooled: Ocular Fellow Eye: Ocular TEAEs are summarized for the fellow eye for all subjects who randomized to sham monthly and sham EOM treatment groups.
  Sham Monthly: Subjects received sham injections once monthly for 12 months.
  Sham EOM: Subjects received sham injections EOM for 12 months. The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
- Pegcetacoplan Monthly: Non-ocular: Non-ocular (systemic) TEAEs are summarized for all subjects who received IVT injections of pegcetacoplan 15 mg/100 μL once monthly for 12 months.
- Pegcetacoplan EOM: Non-ocular: Non-ocular (systemic) TEAEs are summarized for all subjects who received IVT injections of pegcetacoplan 15 mg/100 μL EOM for 12 months.
- Sham Pooled: Non-ocular: Non-ocular (systemic) TEAEs are summarized for all subjects who randomized to sham monthly and sham EOM treatment groups.
  Sham Monthly: Subjects received sham injections once monthly for 12 months.
  Sham EOM: Subjects received sham injections EOM for 12 months. The procedure for sham injection was the same as that used for IVT injection until the actual injection but no actual injection occurred.
Arm/Group | Pegcetacoplan Monthly: Ocular Study Eye | Pegcetacoplan EOM: Ocular Study Eye | Sham Pooled: Ocular Study Eye | Pegcetacoplan Monthly: Ocular Fellow Eye | Pegcetacoplan EOM: Ocular Fellow Eye | Sham Pooled: Ocular Fellow Eye | Pegcetacoplan Monthly: Non-ocular | Pegcetacoplan EOM: Non-ocular | Sham Pooled: Non-ocular
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/79 | 0/81 | 0/86 | 0/79 | 0/81 | 0/86 | 2/79 | 2/81
Serious Adverse Events (participants affected / at risk) | 4/86 | 2/79 | 1/81 | 0/86 | 0/79 | 1/81 | 12/86 | 23/79 | 16/81
Other Adverse Events (participants affected / at risk) | 51/86 | 35/79 | 25/81 | 12/86 | 8/79 | 10/81 | 23/86 | 18/79 | 23/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegcetacoplan Monthly: Ocular Study Eye (N=86) | Pegcetacoplan EOM: Ocular Study Eye (N=79) | Sham Pooled: Ocular Study Eye (N=81) | Pegcetacoplan Monthly: Ocular Fellow Eye (N=86) | Pegcetacoplan EOM: Ocular Fellow Eye (N=79) | Sham Pooled: Ocular Fellow Eye (N=81) | Pegcetacoplan Monthly: Non-ocular (N=86) | Pegcetacoplan EOM: Non-ocular (N=79) | Sham Pooled: Non-ocular (N=81)
Endophthalmitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry age-related macular degeneration (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mitral valve calcification (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epidural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal claudication (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device extrusion (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pegcetacoplan Monthly: Ocular Study Eye (N=86) | Pegcetacoplan EOM: Ocular Study Eye (N=79) | Sham Pooled: Ocular Study Eye (N=81) | Pegcetacoplan Monthly: Ocular Fellow Eye (N=86) | Pegcetacoplan EOM: Ocular Fellow Eye (N=79) | Sham Pooled: Ocular Fellow Eye (N=81) | Pegcetacoplan Monthly: Non-ocular (N=86) | Pegcetacoplan EOM: Non-ocular (N=79) | Sham Pooled: Non-ocular (N=81)
Conjunctival haemorrhage (Eye disorders) | 16 | 9 | 8 | 2 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 19 | 7 | 1 | 4 | 2 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 12 | 3 | 6 | 1 | 1 | 1 | 0 | 0 | 0
Neovascular age-related macular degeneration (Eye disorders) | 10 | 5 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 4 | 9 | 3 | 3 | 4 | 2 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 2 | 4 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 5 | 2 | 3 | 2 | 0 | 2 | 0 | 0 | 0
Dry eye (Eye disorders) | 3 | 1 | 5 | 2 | 1 | 4 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 7 | 8 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 5
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 7
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 8
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT02503332/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT02503332/SAP_001.pdf